CLINICAL TRIAL: NCT07037498
Title: Effects of Moringa Oleifera and Royal Jelly Supplementation on Nutritional Status and Cognitive Function in Adolescent Girls in Takalar District, South Sulawesi, Indonesia: Protocol Study
Brief Title: Effect of Moringa Royal Jelly on the Nutritional Status and Cognitive Level of Adolescent Girls
Acronym: MRJ
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Musfira, Department Nutrition, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2739/UN4.14.1/TP.01.02/2024; Nutrition (Other: Hasanuddin University)
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Undernutrition; Anemia; Stunting; Cognitive Function 1, Social
Keywords: Nutrition
MeSH Terms: conditions — Malnutrition; Anemia; Growth Disorders | interventions — flocculant protein MO 2.1, Moringa oleifera; royal jelly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRJ Supplementation Group (Experimental): Participants in this arm receive MRJ capsules containing 490 mg Moringa oleifera extract and 10 mg royal jelly, taken twice per week for 12 months. The supplementation is accompanied by standardized nutrition education delivered through TikTok videos. Adherence is monitored weekly via teacher-supervised log sheets and WhatsApp documentation.
  Interventions: Dietary Supplement: Moringa Oleifera
- IFA Tablet Group (Control) (Active Comparator): Participants in this arm receive weekly iron-folic acid (IFA) tablets according to national guidelines (60 mg elemental iron and 400 µg folic acid) for 12 months. They also receive the same standardized nutrition education via TikTok videos. Adherence is tracked using weekly log sheets verified by teachers and supported by WhatsApp photo submissions.
  Interventions: Dietary Supplement: Moringa Oleifera

INTERVENTIONS:
Dietary Supplement: Moringa Oleifera — Participants receive MRJ capsules containing 490 mg of Moringa oleifera leaf extract and 10 mg of royal jelly, taken orally twice per week for 12 months. The capsules are plant-based, produced using locally sourced ingredients, and are part of a food-based supplementation strategy developed as an alternative to iron-folic acid tablets. The intervention is combined with standardized nutrition education via TikTok videos. Adherence is monitored weekly through teacher log sheets and WhatsApp documentation. and Participants receive iron-folic acid (IFA) tablets containing 60 mg of elemental iron and 400 µg of folic acid, taken orally once per week for 12 months in accordance with Indonesia's national supplementation guidelines for adolescent girls. This control intervention is combined with the same standardized nutrition education via TikTok videos. Compliance is tracked weekly through teacher-supervised control sheets and WhatsApp photo submissions.
  Other Names: Royal jelly; edukasi

SUMMARY:
The goal of this clinical trial is to learn whether a locally developed supplement called MRJ - a combination of Moringa oleifera (drumstick tree) extract and royal jelly - can improve the nutritional status and cognitive function of adolescent girls more effectively than standard iron and folic acid (IFA) tablets.

The main questions it aims to answer are:

Does MRJ supplementation lead to better improvements in nutrition (e.g., hemoglobin, body measurements)?

Does MRJ supplementation enhance cognitive function compared to IFA tablets?

Researchers will compare MRJ capsules to IFA tablets (the standard of care) among adolescent girls.

Participants will:

Take 2 MRJ capsules per week (intervention group) or 1 IFA tablet per week (control group) for 12 months

Receive nutrition education via short TikTok-based videos

Have their adherence monitored weekly by teachers and through WhatsApp photos

Measurements will be taken at the start, 6 months, and 12 months, including:

Height, weight, and mid-upper arm circumference (MUAC)

Hemoglobin levels via finger-prick blood test

Dietary intake using a 24-hour recall and food frequency questionnaire (FFQ)

Cognitive function assessed with the Culture Fair Intelligence Test (CFIT)

Participants are healthy junior and senior high school girls aged 10-18 years from Galesong Selatan, Takalar District, South Sulawesi, Indonesia.

Potential side effects (e.g., nausea or stomach discomfort) will be monitored according to school health protocols.

The findings may support the use of culturally appropriate, nutrient-rich interventions for improving adolescent girls' health and future well-being.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate whether a locally produced supplement, MRJ (a combination of Moringa oleifera extract and royal jelly), can improve nutritional status and cognitive function among adolescent girls in South Sulawesi, Indonesia, compared to the standard iron and folic acid (IFA) tablets provided by the government. If proven effective, MRJ may serve as a culturally acceptable and nutrient-rich alternative to support adolescent health and development.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 10-19 years (2) Adolescent girls' who are active in grades 1 and 2 (junior high and senior high)

Exclusion Criteria:

* (3) Severe nutritional or health conditions (e.g., severe anemia, severe malnutrition, allergies), determined through clinical histories and validated self-reports.

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 372 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2026-02-17 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index-for-Age Z-score (BMI-for-age) | Baseline, 6 months, and 12 months
  Mean change in BMI-for-age z-scores as per WHO AnthroPlus standards, measured at baseline, 6 months, and 12 months.

SECONDARY OUTCOMES:
Change in Mid-Upper Arm Circumference (MUAC) | Baseline, 6 months, and 12 months
  Mean change in mid-upper arm circumference (cm) measured using standard non-stretchable tape.
Change in cognitive function score (CFIT) | Baseline and 12 months
  Change in cognitive function as assessed using the Culture Fair Intelligence Test (CFIT) at baseline and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Schools under the supervision of Puskesmas Bonto Kassi, Galesong Selatan, Takalar District, South Sulawesi, Indonesia, Takalar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that will be shared include de-identified data on anthropometric measures (BMI-for-age, height-for-age, MUAC), hemoglobin levels, dietary intake (24-hour recall and FFQ), and cognitive function scores (CFIT results). All shared data will be anonymized and stripped of any personal identifiers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified individual participant data (IPD) will be available beginning 6 months after publication of the primary results and will remain available for up to 5 years thereafter.
Access Criteria: Qualified researchers with a scientifically sound proposal may request access to the de-identified data. Access will be granted for purposes of academic research, meta-analysis, or systematic review. Requests should be submitted in writing to the principal investigator or sponsor institution and must include a data use agreement.

REFERENCES:
- [Result] 1. Patton GC, Sawyer SM, Santelli JS, et al. Our future: a Lancet commission on adolescent health and wellbeing. Lancet. 2016;387(10036):2423-78. 2. World Health Organization. Nutrition in adolescence: issues and challenges for the health sector. Geneva: WHO; 2005. 3. Black MM. Micronutrient deficiencies and cognitive functioning. J Nutr. 2003;133(11 Suppl 2):3927S-31S. 4. Best C, Neufingerl N, Van Geel L, van den Briel T, Osendarp S. The nutritional status of school-aged children: why should we care? Food Nutr Bull. 2010;31(3):400-17. 5. UNICEF. The State of the World's Children 2019: Children, food and nutrition. New York: UNICEF; 2019. 6. World Health Organization. Anaemia in women and children. Geneva: WHO; 2023. 7. Health Research and Development Agency. Basic Health Research 2018. Jakarta: Ministry of Health, Republic of Indonesia; 2018. 8. Ministry of Health of the Republic of Indonesia. Indonesia Health Profile 2023. Jakarta: MoH; 2024. 9. Dewey KG, Begum K. Long-term consequences of stunting in early life. Matern Child Nutr. 2011;7(Suppl 3):5-18. 10. Hadju V, Salmah AU, Natsir R, et al. Stunting and its risk factors among adolescent girls in South Sulawesi. Media Gizi Masyarakat Indonesia. 2020;5(2):59-66. 11. Walker SP, Chang SM, Powell CA, et al. Effects of early childhood psychosocial stimulation and nutritional supplementation on cognition and education in growth-stunted Jamaican children. Lancet. 2005;366(9499):1804-7. 12. Grantham-McGregor S, Cheung YB, Cueto S, et al. Developmental potential in the first 5 years for children in developing countries. Lancet. 2007;369(9555):60-70. 13. Prentice AM, Ward KA, Goldberg GR, et al. Critical windows for nutritional interventions against stunting. Am J Clin Nutr. 2013;97(5):911-8. 14. Stoltzfus RJ. Iron deficiency: global prevalence and consequences. Food Nutr Bull. 2003;24(4 Suppl):S99-103. 15. Ministry of Health of the Republic of Indonesia. Indonesia Nutrition Status Survey (SSGI) 2023. Jakarta: MoH; 2024.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT07037498/Prot_SAP_ICF_000.pdf